CLINICAL TRIAL: NCT01994720
Title: A Randomised, Double-Blind, Multinational Study to Prevent Major Vascular Events With Ticagrelor Compared to Aspirin (ASA) in Patients With Acute Ischaemic Stroke or TIA.
Brief Title: [SOCRATES -Acute Stroke Or Transient IsChaemic Attack TReated With Aspirin or Ticagrelor and Patient OutcomES]
Acronym: SOCRATES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D5134C00001; 2012-003895-38 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2013-11-26 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Ischaemic Stroke; Transient Ischaemic Attack
Keywords: Acute ischaemic stroke.; Transient ischaemic attack.
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ticagrelor (Experimental)
  Interventions: Drug: ticagrelor
- Acetylsalicylic acid (ASA) (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid (ASA)

INTERVENTIONS:
Drug: ticagrelor — ticagrelor, 180 mg (two tablets of 90 mg) loading dose on Day 1 followed by 90 mg twice daily.
  Arms: ticagrelor
Drug: Acetylsalicylic acid (ASA) — ASA, 300 mg (three tablets of 100 mg) on Day 1, followed by 100 mg once daily.
  Arms: Acetylsalicylic acid (ASA)

SUMMARY:
The primary objective of the study is to compare the effect of 90-day treatment with ticagrelor (180 mg [two 90 mg tablets] loading dose on Day 1 followed by 90 mg twice daily maintenance dose for the remainder of the study) vs acetylsalicylic acid (ASA)-aspirin (300 mg [three 100 mg tablets] loading dose on Day 1 followed by 100 mg once daily maintenance dose for the remainder of the study) for the prevention of major vascular events (composite of stroke, myocardial infarction [MI], and death) in patients with acute ischaemic stroke or transient ischaemic attack (TIA).

ELIGIBILITY:
Inclusion Criteria:

* Men or women equal or elder 40 years of age
* Either acute ischaemic stroke or high-risk TIA as defined here and randomisation occurring within 24 hours after onset of symptoms

Key Exclusion Criteria:

* Planned use of antithrombotic therapy in addition to study medication including antiplatelets (eg, open label ASA, GPIIb/IIIa inhibitors, clopidogrel, ticlopidine, prasugrel, dipyridamole, ozagrel, cilostazol) and anticoagulants (eg, warfarin, oral thrombin and factor Xa inhibitors, bivalirudin, hirudin, argatroban, unfractionated and low molecular weight heparins). - Any history of atrial fibrillation, ventricular aneurysm or suspicion of cardioembolic pathology for TIA or stroke. - Planned carotid, cerebrovascular, or coronary revascularisation that requires halting study medication within 7 days of randomisation. - Receipt of any intravenous or intra-arterial thrombolysis or mechanical thrombectomy within 24 hours prior to randomisation - History of previous symptomatic non-traumatic intracerebral bleed at any time (asymptomatic microbleeds do not qualify), gastrointestinal (GI) bleed within the past 6 months, or major surgery within 30 days.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13307 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (521):
- United States (115):
  - Research Site, Montgomery, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Fort Smith, Arkansas
  - Research Site, Fullerton, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Newport, California
  - Research Site, Oakland, California
  - Research Site, San Diego, California
  - Research Site, Stanford, California
  - Research Site, Torrance, California
  - Research Site, Englewood, Colorado
  - Research Site, Altamonte Springs, Florida
  - Research Site, Aventura, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Weston, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Glenview, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Alexandria, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, West Bloomfield, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Helena, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Lebanon, New Hampshire
  - Research Site, Bayonne, New Jersey
  - Research Site, Edison, New Jersey
  - Research Site, Englewood, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, West Orange, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Clackamas, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Allentown, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Baytown, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Harlingen, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Southlake, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Martín
- Australia (12):
  - Research Site, Adelaide
  - Research Site, Bedford Park
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Darlinghurst
  - Research Site, Footscray
  - Research Site, Herston
  - Research Site, New Lambton Heights
  - Research Site, Parkville
  - Research Site, Southport
  - Research Site, Sydney
  - Research Site, Woodville
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Assebroek
  - Research Site, Bruges
  - Research Site, Brussels (Woluwé-St-Lambert)
  - Research Site, Ghent
  - Research Site, Godinne
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Tielt
  - Research Site, Wilrijk
- Brazil (8):
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (15):
  - Research Site, Botevgrad
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Lukovit
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sandanski
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Teteven
  - Research Site, Yambol
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (7):
  - Research Site, Concepción
  - Research Site, Los Ángeles
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Temuco
  - Research Site, Valdivia
  - Research Site, Viña del Mar
- China (26):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chongqin
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Huai'an
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhanjiang
- Czechia (10):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Liberec
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Trutnov
- France (24):
  - Research Site, Antony
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Corbeil-Essonnes
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, La Roche-sur-Yon
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Lille
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pringy
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (13):
  - Research Site, Altenburg
  - Research Site, Bad Neustadt an der Saale
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Minden
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Wiesbaden
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Kowloon
  - Research Site, Shatin
- Hungary (12):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron-Balf
  - Research Site, Szekszárd
  - Research Site, Székesfehérvár
- Israel (6):
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (19):
  - Research Site, Carrara
  - Research Site, Città di Castello
  - Research Site, Foligno
  - Research Site, Genova
  - Research Site, Gubbio
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Piacenza
  - Research Site, Pisa
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Siena
  - Research Site, Varese
  - Research Site, Verona
  - Research Site, Vibo Valentia
- Japan (88):
  - Research Site, Aki-gun
  - Research Site, Asahikawa-shi
  - Research Site, Chiba
  - Research Site, Chikushi-gun
  - Research Site, Chikushino-shi
  - Research Site, Chitose-shi
  - Research Site, Daito-shi
  - Research Site, Date-gun
  - Research Site, Eniwa-shi
  - Research Site, Fujinomiya-shi
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Fukuyama-shi
  - Research Site, Gifu
  - Research Site, Hachioji-shi
  - Research Site, Hakodate-shi
  - Research Site, Hamada-shi
  - Research Site, Hanamaki-shi
  - Research Site, Hatsukaichi-shi
  - Research Site, Hidaka-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Higashiosaka-shi
  - Research Site, Hitachi-shi
  - Research Site, Ina-shi
  - Research Site, Itami-shi
  - Research Site, Izumisano
  - Research Site, Izumo-shi
  - Research Site, Kaga-shi
  - Research Site, Kagoshima
  - Research Site, Kakegawa-shi
  - Research Site, Kamakura-shi
  - Research Site, Kashiwazaki-shi
  - Research Site, Kasuga-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Kochi
  - Research Site, Koga-shi
  - Research Site, Komatsu-shi
  - Research Site, Komoro-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Maizuru-shi
  - Research Site, Marugame-shi
  - Research Site, Matsudo-shi
  - Research Site, Matsuyama
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Nakano
  - Research Site, Nakano-shi
  - Research Site, Narita-shi
  - Research Site, Nihonmatsu-shi
  - Research Site, Okayama
  - Research Site, Okinawa-shi
  - Research Site, Onga-gun
  - Research Site, Ookawa-shi
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Sagamihara-shi
  - Research Site, Saijo-shi
  - Research Site, Sakaishi
  - Research Site, Sanuki-shi
  - Research Site, Sapporo
  - Research Site, Sayama-shi
  - Research Site, Sendai
  - Research Site, Shiroishi-shi
  - Research Site, Shizuoka
  - Research Site, Suita-shi
  - Research Site, Suwa-shi
  - Research Site, Tachikawa-shi
  - Research Site, Takasaki-shi
  - Research Site, Takayama-shi
  - Research Site, Tokushima
  - Research Site, Toyama
  - Research Site, Toyohashi
  - Research Site, Toyota-shi
  - Research Site, Tsu
  - Research Site, Ube-shi
  - Research Site, Ueda-shi
  - Research Site, Uji-shi
  - Research Site, Ureshino-shi
  - Research Site, Utsunomiya
  - Research Site, Yokohama
  - Research Site, Zentsuji-shi
- Mexico (6):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Del. Cuauhtemoc
  - Research Site, Distrito Federal
  - Research Site, Monterrey
- Peru (4):
  - Research Site, Bellavista
  - Research Site, Callao
  - Research Site, Cusco
  - Research Site, Lima
- Philippines (8):
  - Research Site, Baguio City
  - Research Site, Cagayan de Oro
  - Research Site, Cebu
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Pasay
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (16):
  - Research Site, Bialystok
  - Research Site, Chełm
  - Research Site, Działdowo
  - Research Site, Gdansk
  - Research Site, Gmina Końskie
  - Research Site, Gryfice
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Ostrołęka
  - Research Site, Sandomierz
  - Research Site, Warsaw
  - Research Site, Włocławek
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Sibiu
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (16):
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Ufa
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (6):
  - Research Site, Levoča
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Spišská Nová Ves
  - Research Site, Trnava
  - Research Site, Žilina
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (11):
  - Research Site, Albacete
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Santiago(A Coruña)
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
- Sweden (13):
  - Research Site, Falun
  - Research Site, Gothenburg
  - Research Site, Halmstad
  - Research Site, Karlstad
  - Research Site, Lidköping
  - Research Site, Linköping
  - Research Site, Malmo
  - Research Site, Mora
  - Research Site, Norrköping
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västerås
- Switzerland (10):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Chur
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Sankt Gallen
  - Research Site, Villars-sur-Glâne
  - Research Site, Zurich
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan Hsien
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chon Buri
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Patumthani
  - Research Site, Rajthevi
  - Research Site, Ratchathewi
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya
- Ukraine (8):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Diener HC, Easton JD, Hart RG, Kasner S, Kamel H, Ntaios G. Review and update of the concept of embolic stroke of undetermined source. Nat Rev Neurol. 2022 Aug;18(8):455-465. doi: 10.1038/s41582-022-00663-4. Epub 2022 May 10. PMID 35538232
- [Derived] Evans SR, Knutsson M, Amarenco P, Albers GW, Bath PM, Denison H, Ladenvall P, Jonasson J, Easton JD, Minematsu K, Molina CA, Wang Y, Wong KL, Johnston SC. Methodologies for pragmatic and efficient assessment of benefits and harms: Application to the SOCRATES trial. Clin Trials. 2020 Dec;17(6):617-626. doi: 10.1177/1740774520941441. Epub 2020 Jul 15. PMID 32666831
- [Derived] Cucchiara B, George DK, Kasner SE, Knutsson M, Denison H, Ladenvall P, Amarenco P, Johnston SC. Disability after minor stroke and TIA: A secondary analysis of the SOCRATES trial. Neurology. 2019 Aug 13;93(7):e708-e716. doi: 10.1212/WNL.0000000000007936. Epub 2019 Jul 11. PMID 31296654
- [Derived] Easton JD, Denison H, Evans SR, Knutsson M, Amarenco P, Albers GW, Ladenvall P, Minematsu K, Molina CA, Wang Y, Wong KL, Johnston SC; SOCRATES Steering Committee and Investigators. Estimated treatment effect of ticagrelor versus aspirin by investigator-assessed events compared with judgement by an independent event adjudication committee in the SOCRATES trial. Int J Stroke. 2019 Dec;14(9):908-914. doi: 10.1177/1747493019851282. Epub 2019 May 15. PMID 31092152
- [Derived] Molina CA, Johnston SC, Ladenvall P, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Knutsson M, Minematsu K, Rother J, Wang Y, Wong KSL; SOCRATES Steering Committee and Investigators. Time to Loading Dose and Risk of Recurrent Events in the SOCRATES Trial. Stroke. 2019 Mar;50(3):675-682. doi: 10.1161/STROKEAHA.118.022675. PMID 30776996
- [Derived] Wong KSL, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Himmelmann A, Kasner SE, Knutsson M, Ladenvall P, Minematsu K, Molina CA, Wang Y, Johnston SC; SOCRATES Steering Committee and Investigators. Efficacy and Safety of Ticagrelor in Relation to Aspirin Use Within the Week Before Randomization in the SOCRATES Trial. Stroke. 2018 Jul;49(7):1678-1685. doi: 10.1161/STROKEAHA.118.020553. Epub 2018 Jun 18. PMID 29915123
- [Derived] Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Hill MD, Jonasson J, Kasner SE, Ladenvall P, Minematsu K, Molina CA, Wang Y, Wong KSL, Johnston SC; SOCRATES Steering Committee and Investigators. Ticagrelor Versus Aspirin in Acute Embolic Stroke of Undetermined Source. Stroke. 2017 Sep;48(9):2480-2487. doi: 10.1161/STROKEAHA.117.017217. Epub 2017 Jul 18. PMID 28720658
- [Derived] Easton JD, Aunes M, Albers GW, Amarenco P, Bokelund-Singh S, Denison H, Evans SR, Held P, Jahreskog M, Jonasson J, Minematsu K, Molina CA, Wang Y, Wong KSL, Johnston SC; SOCRATES Steering Committee and Investigators. Risk for Major Bleeding in Patients Receiving Ticagrelor Compared With Aspirin After Transient Ischemic Attack or Acute Ischemic Stroke in the SOCRATES Study (Acute Stroke or Transient Ischemic Attack Treated With Aspirin or Ticagrelor and Patient Outcomes). Circulation. 2017 Sep 5;136(10):907-916. doi: 10.1161/CIRCULATIONAHA.117.028566. Epub 2017 Jun 27. PMID 28655834
- [Derived] Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Hill MD, Jonasson J, Kasner SE, Ladenvall P, Minematsu K, Molina CA, Wang Y, Wong KSL, Johnston SC; SOCRATES Steering Committee and Investigators. Efficacy and safety of ticagrelor versus aspirin in acute stroke or transient ischaemic attack of atherosclerotic origin: a subgroup analysis of SOCRATES, a randomised, double-blind, controlled trial. Lancet Neurol. 2017 Apr;16(4):301-310. doi: 10.1016/S1474-4422(17)30038-8. Epub 2017 Feb 23. PMID 28238711
- [Derived] Wang Y, Minematsu K, Wong KS, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Jonasson J, Molina CA, Johnston SC; SOCRATES Steering Committee and Investigators. Ticagrelor in Acute Stroke or Transient Ischemic Attack in Asian Patients: From the SOCRATES Trial (Acute Stroke or Transient Ischemic Attack Treated With Aspirin or Ticagrelor and Patient Outcomes). Stroke. 2017 Jan;48(1):167-173. doi: 10.1161/STROKEAHA.116.014891. Epub 2016 Nov 29. PMID 27899747
- [Derived] Held P, Himmelmann A, Ditmarsch M. Ticagrelor for the treatment of atherosclerotic disease: insights from the PARTHENON clinical development program. Future Cardiol. 2016 Jul;12(4):405-18. doi: 10.2217/fca-2016-0028. Epub 2016 May 10. PMID 27160944
- [Derived] Johnston SC, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Jonasson J, Minematsu K, Molina CA, Wang Y, Wong KS; SOCRATES Steering Committee and Investigators. Ticagrelor versus Aspirin in Acute Stroke or Transient Ischemic Attack. N Engl J Med. 2016 Jul 7;375(1):35-43. doi: 10.1056/NEJMoa1603060. Epub 2016 May 10. PMID 27160892
- See also: CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1836&filename=d5134c00001-revised-csp-2-redacted_1July2015.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 13307 patients were enrolled from 674 study sites in 33 countries. The first patient was enrolled on 07 January 2014. The last patient visit took place on 02 March 2016.
Pre-assignment Details: Enrolled patients randomised to study drug: 99.2%; n=13199 Patients who were not randomised: 0.8%; n=108 Patients with eligibility criteria not fulfilled: 0.7%; n=93 Patient decision: 0.1%; n=15
Groups:
- Ticagrelor 90 mg: Ticagrelor 90 mg twice daily (BD)
- ASA 100 mg: ASA 100 mg once daily (OD)
Period: Overall Study
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Started | 6589 | 6610
Completed | 6543 (Includes patients who did not withdraw informed consent prior to the Study Closure Visit) | 6554 (Includes patients who did not withdraw informed consent prior to the Study Closure Visit)
Not Completed | 46 | 56
Not completed — Withdrawal by Subject | 46 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 90 mg | ASA 100 mg | Total
Number analyzed (Participants) | 6589 | 6610 | 13199
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (11.23) | 65.9 (11.37) | 65.9 (11.30)
Age, Customized [Number; unit: Participants]
  <65 years | 3021 | 3007 | 6028
  Between 65 and 75 years | 2064 | 2112 | 4176
  >75 years | 1504 | 1491 | 2995
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2759 | 2724 | 5483
  Male | 3830 | 3886 | 7716
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 566 | 558 | 1124
  Not Hispanic or Latino | 6023 | 6050 | 12073
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 69 | 74 | 143
  Asian | 1957 | 1949 | 3906
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 119 | 120 | 239
  White | 4374 | 4410 | 8784
  Other | 66 | 56 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Stroke/MI/Death
Description: Participants with stroke, MI or death. If no event, censoring occures at the minimum of (last date of event assessment, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 442 | 497
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Composite of stroke/MI/death; Test type: Superiority or Other; p = 0.0670, Regression, Cox — In order to address the issue of multiple testing, a hierarchical test sequence will be used. Tested at 4.98% level; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.78 to 1.01]

2. Secondary Outcome: Number of Participants With Ischaemic Stroke
Description: Participants with ischaemic stroke. If no event, censoring occures at the minimum of (last date of event assessment, date of death, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 385 | 441
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Ischemic stroke; Test type: Superiority or Other; p = 0.0462, Regression, Cox — If the treatment effect on the primary efficacy variable is significant at the 4.98% level, the secondary efficacy variable will be tested in a confirmatory sense. Otherwise it will be tested in an exploratory manner; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.76 to 1.00]

3. Secondary Outcome: Net Clinical Outcome
Description: Participants with stroke, MI, death or life-threatening bleeding. If no event, censoring occures at the minimum of (last date of event assessment, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 457 | 508
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.0928, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.79 to 1.02]

4. Secondary Outcome: Number of Participants With Composite of Ischaemic Stroke, MI and CV Death
Description: Participants with ischaemic stroke, MI or CV death. If no event, censoring at the minimum of (last date of event assessment, date of death from non-CV causes, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 423 | 475
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.0771, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.78 to 1.01]

5. Secondary Outcome: Number of Participants With All-Cause Death
Description: Participants with all-cause death. If no event, censoring at the minimum of (last date of event assessment, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 68 | 58
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.3641, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.83 to 1.67]

6. Secondary Outcome: Number of Participants With CV Death
Description: Participants with CV death. If no event, censoring at the minimum of (last date of event assessment, date of death from non-CV causes, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 41 | 35
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.4828, Regression, Cox; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.75 to 1.85]

7. Secondary Outcome: Number of Participants With MI
Description: Participants with MI. If no event, censoring at the minimum of (last date of event assessment, date of death, end of treatment date, day 97)
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 25 | 21
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.5457, Regression, Cox; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.67 to 2.14]

8. Secondary Outcome: Number of Participants by Severity of Stroke and Overall Disability
Description: Analysis of severity of stroke and overall disability of patients, using the modified Rankin Score, mRS.
  Modified Rankin Score:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
  Disability defined as mRS > 1.
  Odds ratio and p-value are calculated for ticagrelor versus ASA from a logistic regression model with treatment group, history of stroke and NIHSS (National Institutes of Health Stroke Scale) at baseline as explanatory variables.
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 1107 | 1194
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.1393, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.85 to 1.02]

9. Secondary Outcome: Number of Participants With Stroke
Description: Participants with stroke. If no event, censoring at the minimum of (last date of event assessment, date of death, end of treatment date, day 97)
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 390 | 450
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.0342, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.75 to 0.99]

10. Secondary Outcome: Number of Participants With Fatal Stroke
Description: Participants with fatal stroke. If no event, censoring at the minimum of (last date of event assessment, date of death from non-CV causes, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 18 | 17
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.8557, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.55 to 2.06]

11. Secondary Outcome: Number of Participants With Disabling Stroke
Description: Participants with disabling stroke. If no event, censoring at the minimum of (last date of event assessment, date of death, end of treatment date, day 97).
Time Frame: From randomization up to 97 days
Population: The population was the full analysis set, which included all randomized patients.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6589 | 6610
Participants | 277 | 307
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p = 0.2126, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.77 to 1.06]

12. Secondary Outcome: Change in NIHSS
Description: Change from baseline to end of treatment visit in NIHSS (National Institutes of Health Stroke Scale):
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke.
Time Frame: From randomization up to 97 days
Population: NIHSS in patients with an index stroke event
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 4798 | 4869
Participants
  <=-5 | 132 | 127
  -4 | 403 | 438
  -3 | 779 | 810
  -2 | 1088 | 1073
  -1 | 1099 | 1131
  0 | 681 | 683
  1 | 67 | 79
  2 | 28 | 31
  3 | 18 | 16
  4 | 13 | 11
  5 | 6 | 6
  >5 | 10 | 14
  Missing | 474 | 450

13. Secondary Outcome: EQ-5D at Visit 1 (Enrolment)
Description: EQ-5D (EuroQol five dimensions questionnaire) index score using the UK tariff.
  EQ-5D is a self assessment of 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. For each dimension responders are asked to state their status on a three level ordinal scale; whether they experience no problems (Level 1), some problems (Level 2) or severe problems (Level 3). Health states defined by the 5 dimensions can be converted into a weighted health state index (health state utility) by applying scores from the EQ-5D value sets elicited from general population samples.
  The higher the index score the better the health state. In this study index scores ran from -0.59 to 1.
Time Frame: Visit 1 (Enrolment)
Population: Include only results from patients who visit the site in-person.
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6497 | 6512
Index score | 0.70 (0.297) | 0.70 (0.298)

14. Secondary Outcome: EQ-5D at Visit 2 (Day 7+-2d)
Description: as for outcome 13
Time Frame: Visit 2 (Day 7+-2d)
Population: Include only results from patients who visit the site in-person.
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 5883 | 5909
Index score | 0.80 (0.244) | 0.79 (0.262)

15. Secondary Outcome: EQ-5D (EuroQol Five Dimensions Questionnaire) at End of Treatment Visit
Description: EQ-5D index score using the UK tariff.
  EQ-5D is a self assessment of 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. For each dimension responders are asked to state their status on a three level ordinal scale; whether they experience no problems (Level 1), some problems (Level 2) or severe problems (Level 3). Health states defined by the 5 dimensions can be converted into a weighted health state index (health state utility) by applying scores from the EQ-5D value sets elicited from general population samples.
  The higher the index score the better the health state. In this study index scores ran from -0.59 to 1.
Time Frame: End of treatment visit (Day 90+-7d)
Population: Include only results from patients who visit the site in-person.
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 5817 | 5893
Index score | 0.85 (0.203) | 0.84 (0.208)

16. Secondary Outcome: EQ-5D (EuroQol Five Dimensions Questionnaire) at Premature Treatment Discontinuation Visit
Description: as for outcome 15
Time Frame: Premature treatment discontinuation visit(<15 days after last dose)
Population: Include only results from patients who visit the site in-person. The Premature Treatment Discontinuation visit (PTDV) is only done for patients who prematurely and permanently stop study medication.
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 787 | 633
Index score | 0.72 (0.330) | 0.68 (0.364)

17. Secondary Outcome: Number of Participants With PLATO Major Bleeding Event
Description: Participants with PLATO Major bleeding. If no event, censoring occures at the minimum of (last date of event assessment, date of death, end of treatment date, day 97).
  PLATO Major bleeding is defined as a bleed that is any one of:
  * Fatal
  * Intracranial (excluding asymptomatic haemorrhagic transformations of ischemic brain infarctions and excluding micro-hemorrhages <10 mm evident only on gradient-echo MRI)
  * Intrapericardial bleed with cardiac tamponade
  * Hypovolaemic shock or severe hypotension due to bleeding and requiring pressors or surgery
  * Significantly disabling (eg. intraocular with permanent vision loss)
  * Clinically overt or apparent bleeding associated with a decrease in Hb of more than 30 g/L (1.9 mmol/L; 0.465 mmol/L)
  * Transfusion of 2 or more units (whole blood or packed red blood cells [PRBCs]) for bleeding.
Time Frame: From randomization up to 97 days
Population: The population was the safety analysis set, which included all patients who received at least 1 dose of randomized ticagrelor or ASA and for whom post-dose data are available.
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6549 | 6581
Participants | 31 | 38
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; PLATO Major bleeding; Test type: Superiority or Other; p = 0.4511, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.52 to 1.34]

18. Secondary Outcome: Number of Participants With Premature Discontinuation of Study Drug Due to Any Bleeding Adverse Event
Description: Participants discontinuation of study drug due to any bleeding adverse event. If no event, censoring occures at the minimum of (last date of event assessment, date of death, end of treatment date, day 97).
Time Frame: Time from first dose and up to and including 7 days following the date of last dose of the study
Population: as for outcome 17
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 90 mg | ASA 100 mg
Number analyzed (Participants) | 6549 | 6581
Participants | 82 | 37
Statistical Analysis 1: Comparison: Ticagrelor 90 mg vs ASA 100 mg; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 2.26, 95% CI 2-sided [1.53 to 3.34]

ADVERSE EVENTS:
Time Frame: On or after the date of first dose and up to and including 7 days following the date of last dose of study medication. 97 days if the participant completed treatment according to the study plan.
Description: The population was the safety analysis set, which included all patients who received at least 1 dose of randomized ticagrelor or ASA and for whom post-dose data are available.
  These patients totaled 6549 for ticagrelor and 6581 for ASA.
Groups:
- ASA 100mg: ASA 100 mg once daily (OD)
- Ticagrelor 90mg: Ticagrelor 90 mg twice daily (BD)
Arm/Group | ASA 100mg | Ticagrelor 90mg
Serious Adverse Events (participants affected / at risk) | 533/6581 | 532/6549
Other Adverse Events (participants affected / at risk) | 85/6581 | 383/6549
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA 100mg (N=6581) | Ticagrelor 90mg (N=6549)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 3 (3)
Angina unstable (Cardiac disorders) | 4 (4) | 11 (11)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 21 (21) | 24 (25)
Atrial flutter (Cardiac disorders) | 1 (1) | 3 (3)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 6 (6)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 7 (7) | 7 (7)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 2 (2)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 4 (4)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac mass (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 4 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular asystole (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 6 (6) | 3 (3)
Deafness permanent (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 4 (5) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Intraocular haematoma (Eye disorders) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 7 (8) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 3 (3)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatocellular injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 5 (5) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 2 (2)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otosalpingitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 23 (25) | 19 (19)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subdural empyema (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 8 (8)
Urosepsis (Infections and infestations) | 0 (0) | 4 (4)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Nerve root injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Cardiac function test abnormal (Investigations) | 1 (1) | 0 (0)
Flavivirus test positive (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Extraskeletal myxoid chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (2) | 2 (2)
Basilar artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Capsular warning syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 2 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 27 (27) | 28 (28)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral amyloid angiopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Clumsiness (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 6 (6)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (3) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 4 (5)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 4 (4) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 4 (5) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Internal carotid artery kinking (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 7 (7) | 5 (5)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Meningeal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 2 (2)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Neurodegenerative disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neurological decompensation (Nervous system disorders) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Partial seizures (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 6 (6)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 68 (74) | 55 (57)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 5 (5) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1)
Somatoform disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 6 (6)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 5 (5) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Malacoplakia vesicae (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Platypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (2)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (3)
Haemorrhagic infarction (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (11) | 12 (13)
Hypertensive crisis (Vascular disorders) | 7 (7) | 7 (7)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0)
Subclavian artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASA 100mg (N=6581) | Ticagrelor 90mg (N=6549)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 85 (86) | 383 (425)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No